CLINICAL TRIAL: NCT01841502
Title: The ROLE of ParoXetine in Patients Taking Telaprevir-based Hepatitis C Therapy: Lack of a Drug-drug Interaction? (ROLEX)
Brief Title: Interaction Between Paroxetine and Telaprevir
Acronym: ROLEX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Telaprevir will not be used in NL, no more inclusions are expected.
Sponsor: Radboud University Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AKF UMCN 12.02
Record Dates: First submitted 2013-04-02; First posted 2013-04-26 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis C Infection; Depression
Keywords: telaprevir; paroxetine; interaction; pharmacokinetics
MeSH Terms: conditions — Hepatitis C; Depression | interventions — Paroxetine; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paroxetine alone (Active Comparator): paroxetine 20 mg tablet once daily oral
  Interventions: Drug: Paroxetine
- paroxetine + telaprevir (Experimental): paroxetine 20 mg tablet once daily + telaprevir 1125 mg (3 tablets 375mg) twice daily oral
  Interventions: Drug: Paroxetine; Drug: telaprevir

INTERVENTIONS:
Drug: Paroxetine — paroxetine 20 mg once daily
Drug: telaprevir — telaprevir 1125 mg twice daily
  Arms: paroxetine + telaprevir

SUMMARY:
Hepatitis C (HCV) infected patients are often in need for an antidepressant. The introduction of Direct Acting Antivirals such as telaprevir has greatly improved treatment outcome of HCV infected patients.Telaprevir has been studied with one antidepressant, escitalopram: plasma concentrations of the antidepressant were reduced by 35% and without dose adjustment this may lead to inadequate treatment of depressive symptoms. There is a need for more data on telaprevir drug interactions with other antidepressants.

For a number of reasons, paroxetine may be a good candidate for use together with telaprevir-containing HCV treatment.

The interaction between paroxetine and telaprevir has not been studied before.

DETAILED DESCRIPTION:
HCV infected patients are often in need for an antidepressant. Inadequate treatment of depression during HCV treatment has a negative effect on adherence to HCV treatment, with suboptimal response as a potential result.

The introduction of Direct Acting Antivirals such as telaprevir has greatly improved treatment outcome of HCV infected patients. Telaprevir, however, causes some significant drug-drug interactions and hence co-administration of other medications should preferably only be done based on clinical evidence that such a combination is safe.

Telaprevir has been studied with one antidepressant, escitalopram: plasma concentrations of the antidepressant were reduced by 35% and without dose adjustment this may lead to inadequate treatment of depressive symptoms. Dose titration of escitalopram may be needed but it may take several weeks before a patient has reached a therapeutic dose.

There is a need for more data on telaprevir drug interactions with other antidepressants. First, the data above show that a negative interaction occurs with escitalopram and dose-titration of the antidepressant may take too long to prevent the (re-)occurrence of depressive symptoms. Second, not all patients benefit from escitalopram and those with (prior) treatment failure on escitalopram may require an alternative agent. Third, although escitalopram is generally well-tolerated, side effects may occur and necessitate treatment discontinuation. Finally, especially in the previous intravenous drug users on methadone, escitalopram might not be the antidepressant of choice, since escitalopram as well as methadone are drugs that can lead to QTc interval prolongation and have a risk of Torsades de Pointes.

For a number of reasons, paroxetine may be a good candidate for use together with telaprevir-containing HCV treatment. First, paroxetine has been shown to prevent depressive symptoms in patients initiating HCV treatment with elevated depressive symptoms at baseline. Second, paroxetine is an inhibitor of and is metabolized by CYP2D6 while telaprevir is an inhibitor of and is metabolized by CYP3A, and therefore no drug-drug interaction is expected. Third, paroxetine is one of the most widely prescribed antidepressants with a well-established efficacy and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 65 years at screening.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject has a chronic HCV infection with genotype 1.
* Subject is eligible for telaprevir containing HCV treatment.
* Subject is on a stable dose of 20 mg paroxetine once daily for at least 4 weeks.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Pregnant female (as confirmed by a human chorionic gonadotropin (HCG) test performed less than 6 weeks before Day -1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose of telaprevir.
* Use of relevant concomitant medication, as assessed by a hospital pharmacist (member of the study team).
* Hemoglobin < 12 g/dL (females) or < 13 g/dL (males) (7.4 respectively 8.0 mM).
* Poor- or ultrarapid metabolizer CYP2D6 (based on genetic testing)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
paroxetine area under the curve (AUC) | day -1 and day 14
  paroxetine AUC will be compared intrasubject: day 14 + telaprevir / day -1 (without telaprevir)

SECONDARY OUTCOMES:
paroxetine Cmax and C24 | Day -1 and Day 14
  Comparison of Cmax and C24 of paroxetine intrasubject. Day 14 (+telaprevir) / Day -1 (without telaprevir)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day -1 to Day 28
  Adverse events will be scored during the study
short term HCV RNA response | week 4
  At week 4 HCV RNA will be determined
telaprevir area under the curve (AUC) | Day 14
  Telaprevir pharmacokinetics (PK) will be determined with paroxetine concomitant use. To be compared to historical data

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (7):
- Netherlands (7):
  - Academic Medical Centre Amsterdam, Amsterdam
  - GGD Amsterdam, Amsterdam
  - Reinier de Graaf Groep, Delft
  - University Medical Centre Groningen, Groningen
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Maasstadziekenhuis, Rotterdam
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- See also: dissertation page 185-192 — https://repository.ubn.ru.nl/handle/2066/142579